CLINICAL TRIAL: NCT05839444
Title: A Pilot Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Study to Evaluate the Safety and Tolerability of BioPB-01 in Healthy Adults
Brief Title: A Clinical Study to Evaluate the Safety and Tolerability of BioPB-01 in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BT/220901/PM/SAT
Record Dates: First submitted 2023-03-23; First posted 2023-05-03 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel-group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Stratified block randomization, Sequentially numbered, sealed, opaque envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioPB-01 (Active Comparator): 2 sachets/day, one to be taken orally with (4±1 mins prior) at breakfast and one (4±1 mins prior) at dinner.
  Interventions: Other: BioPB-01
- Placebo (Placebo Comparator): 2 sachets/day, one to be taken orally with (4±1 mins prior) at breakfast and one (4±1 mins prior) at dinner.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: BioPB-01 — 2 sachets/day, one to be taken orally with (4±1 mins prior) at breakfast and one (4±1 mins prior) at dinner
  Arms: BioPB-01
Other: Placebo — 2 sachets/day, one to be taken orally with (4±1 mins prior) at breakfast and one (4±1 mins prior) at dinner
  Arms: Placebo

SUMMARY:
The present study is a randomized, placebo-controlled, parallel-group, double-blind clinical study. Seventy-eight individuals will be screened, and considering a screening failure rate of 20%, approximately 64 participants will be randomized in a ratio of 1:1 to receive either BioPB-01 or Placebo

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are 25 to 55 years of age (inclusive) at the time ofsigning the informed consent form.
2. Participants having good general health (no active or uncontrolled diseases, infections, or conditions).
3. BMI within the range of 24.9 to 34.9 kg/m2 (inclusive).
4. Random blood glucose level <140 mg/dL.
5. Concurrent metformin use is acceptable for indications other than diabetes. (However, the subject and investigator must not change metformin dosing during the three weeks of the study).
6. Non-pregnant and non-lactating females of childbearing potential who agree to use adequate contraception/sexual abstinence throughout the study period.
7. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.
8. Individuals with access to a digital device to fill out the questionnaires.

Exclusion Criteria:

1. Participant has a history of uncontrolled hypertension (i.e., ≥150 mmHg systolic and/or ≥110 mmHg diastolic).
2. Participant with history of post-prandial hypoglycemia (occurring 2-5 hours after food intake) of unknown cause.
3. Abnormal thyroid-stimulating hormone (TSH) levels (<0.4 or > 4.2 μIU/ml).
4. Known case of Type 1 or 2 diabetes.
5. Participant has a history of heart disease and/or cardiovascular disease, kidney disease (dialysis or renal failure), and/or hepatic impairment or disease.
6. Participant has a history of previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the year prior to screening, immune disorder (i.e., HIV/AIDS), or a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to the screening visit.
7. Received a vaccine for COVID-19 or any other vaccination in the 2 weeks prior to screening or planned during the study period, currentCOVID-19 infections, or currently have the post COVID-19 condition as defined by the World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis).
8. Have a known intolerance, sensitivity, or allergy to any of the study products, their ingredients, or any excipients used in the formulation.
9. Individuals who have a known history of diverticulitis.
10. Have a known intolerance, sensitivity, or allergy to milk or soy.
11. Any condition or abnormality that, in the opinion of the Investigator, would compromise the safety of the participant or the quality of the study data.
12. Currently taking dietary supplements other than vitamins and minerals.
13. Taking any other prescription medication at the time of randomization that is known to impact blood sugar and or blood sugar metabolism, as per the Principal Investigator's (PI) discretion.
14. History of smoking, alcohol (heavy drinking as defined by NIAAA [National Institute on Alcohol Abuse and Alcoholism], USA), or substance abuse in the 12 months prior to screening.
15. Receipt or use of an investigational product in another research study within 30 days prior to baseline/Visit 2.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  The gastrointestinal (GI) health assessed using a modified Gastrointestinal Symptom Questionnaire (GSQ) compared to baseline and placebo
To evaluate the safety of 21 days of BioPB-01 administration on | Day 14
  The gastrointestinal (GI) health assessed using a modified Gastrointestinal Symptom Questionnaire (GSQ) compared to baseline and placebo
To evaluate the safety of 21 days of BioPB-01 administration on | Day 7
  The gastrointestinal (GI) health assessed using a modified Gastrointestinal Symptom Questionnaire (GSQ) compared to baseline and placebo
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  Stool consistency using Bristol stool form scale (BSFS) compared to baseline and placebo.This scale is a 7 point ordinal scale of stool types. The participants will be asked to rate their stool consistency and frequency daily to assess abnormal stools, defined as alteration in the frequency or consistency type 1, 2, 6, or 7.
To evaluate the safety of 21 days of BioPB-01 administration on | Day 14
  Stool consistency using Bristol stool form scale (BSFS) compared to baseline and placebo. The participants will be asked to rate their stool consistency and frequency daily to assess abnormal stools, defined as alteration in the frequency or consistency type 1, 2, 6, or 7.
To evaluate the safety of 21 days of BioPB-01 administration on | Day 7
  Stool consistency using Bristol stool form scale (BSFS) compared to baseline and placebo. The participants will be asked to rate their stool consistency and frequency daily to assess abnormal stools, defined as alteration in the frequency or consistency type 1, 2, 6, or 7.
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  Liver function biomarkers Alanine transaminase (ALT)
  Reference range:
  Females: 9-52 U/L Males: 21-72 U/L
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  Liver function biomarkers Aspartate aminotransferase (AST)
  Reference range:
  Females: 14-36 U/L Males: 17-59 U/L
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  Renal function biomarker blood urea nitrogen (BUN) - Female: 7-17 mg/dL or 2.5-6.1 mmol/L Male: 9-20 mg/dL or 3.2-7.1 mmol/L
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  Renal function biomarker Creatinine Reference range: Female: 0.52-1.04 mg/dL or 46-92 μmol/L Male: 0.66-1.25 mg/dL or 58-110 μmol/L
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  Serum electrolytes (sodium) : 137-145 mmol/L
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  Serum electrolytes (potassium): 3.5-5.1 mmol/L
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  Vitals - Blood pressure : Both Systolic and Diastolic pressure will be measured
To evaluate the safety of 21 days of BioPB-01 administration on | Day 21
  Vitals - Pulse rate
To evaluate the safety of 21 days of BioPB-01 administration on | Throughout the study (an average of 21 days)
  The number and percentage of participants having adverse product reaction (as per CTCAE V5.0)

SECONDARY OUTCOMES:
To evaluate the efficacy of BioPB-01 after 21 days of administration by assessing the metabolic health | Day 21
  As assessed by the serum lipid profile (Triglycerides (TG), Total cholesterol (TC), low-density lipoprotein (LDL), and high-density lipoprotein (HDL)) level from Baseline
To evaluate the efficacy of BioPB-01 after 21 days of administration by assessing | Day 21
  The insulin sensitivity as assessed by HOMA-IR from baseline
To evaluate the efficacy of BioPB-01 after 21 days of administration by assessing | Day 21
  The post-prandial insulin response by net incremental area-under-the-curve (AUC) for post-prandial glucose and insulin (30, 60, 90, and 120 min. after standardised meal) from baseline.
To evaluate the efficacy of BioPB-01 after 21 days of administration by assessing | Day 21
  Inflammation by serum C-reactive protein (CRP) level from Baseline
To evaluate the efficacy of BioPB-01 after 21 days of administration by assessing | Day 21
  Satiety using the Appetite/Satiety - using Visual Analog Scale (VAS) from Baseline.
  The scale comprises of 4 main domains: 1) Hunger, 2) Fullness after meals, 3) Thoughts of food, 4) Cravings. The appetite will be analysed based on these four domains on a 100 mm VAS. Reduction in scores as compared to day 0 and placebo will indicate improvement in the appetite/satiety and efficacy of the IP on the appetite/satiety.
To evaluate the efficacy of BioPB-01 after 21 days of administration by assessing | Day 21
  Body weight from baseline.
To evaluate the efficacy of BioPB-01 after 21 days of administration by assessing Fecal short chain fatty acids (SCFA) | Day 21
  Namely acetate, propionate, and butyrate from Baseline. The samples will be analysed using liquid chromatography tandem mass spectrometry (LC-MS/MS).

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Aman Hospital and Research Center, Vadodara, Gujarat
  - Lifecare Hospital, Nashik, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided